CLINICAL TRIAL: NCT07135791
Title: Real-Time Monitoring of Fatigue In Daily Life Among Adults With Cerebral Palsy or Acquired Brain Injury: An Observational Study
Brief Title: Monitoring Fatigue In Daily Life In Adults With Cerebral Palsy or Acquired Brain Injury
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Center for Rehabilitation of Brain Injury (Center for Hjerneskade) (Unknown); Vejlefjord Rehabilitation (Other); Elsass Foundation (Other)
Responsible Party: Principal Investigator, Frederik Dornonville de la Cour, Postdoc, Rigshospitalet, Denmark
Other Study IDs: p-2023-14839
Record Dates: First submitted 2025-07-29; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Fatigue Symptom; Fatigue Intensity; Cerebral Palsy (CP); Acquired Brain Injury Including Stroke; Fatigue, Mental; Fatigue
Keywords: Cerebral palsy; Acquired brain injury; ecological momentary assessment; experience sampling method; real-time monitoring; Fatigue; Real-time fatigue
MeSH Terms: conditions — Fatigue; Cerebral Palsy; Mental Fatigue; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cerebral palsy: Adults with cerebral palsy
  Interventions: Diagnostic Test: Real-time monitoring
- Acquired brain injury: Adults with acquired brain injury
  Interventions: Diagnostic Test: Real-time monitoring
- Healthy volunteers: Adults without neurological conditions
  Interventions: Diagnostic Test: Real-time monitoring

INTERVENTIONS:
Diagnostic Test: Real-time monitoring — Complete a brief 20-item survey 10 times a day for seven consecutive days, while wearing an accelerometer and completing daily sleep diaries.
  Other Names: Ecological Momentary Assessment; Ambulatory assessment

SUMMARY:
The goal of this observational study is to learn about levels and patterns of fatigue in adults with cerebral palsy (CP) and acquired brain injury (ABI) in daily life.

The main question it aims to answer is: How do adults with CP and ABI experience fatigue in daily life?

Researchers will compare data from CP and ABI with healthy volunteers to see if they experience fatigue differently.

Participants will:

* Monitor their symptoms, mood, and behavior in real-time by completing a brief survey on their mobile phone 10 times a day for seven consecutive days.
* Attend a briefing session the day prior to the seven-day period of real-time monitoring.
* Wear an accelerometer for the seven-day period.
* Complete a daily sleep diary for the seven-day period.
* Receive feedback on their real-time monitoring data, sleep and activity data.

DETAILED DESCRIPTION:
Fatigue is a major problem for adults with cerebral palsy (CP) or acquired brain injury (ABI), and contributes to disability, loss of productivity, and poor quality of life.

Qualitative research indicates that fatigue symptoms are dynamic and context-dependent, and the severity of symptoms can fluctuate throughout the day and from day to day.

People living with fatigue may tire more easily, in response to physical or mental exertion, than people without fatigue. Symptoms of fatigue may worsen dramatically and unexpectedly from one moment to the next. It can be very difficult for people to figure out, why they are suddenly overwhelmed by fatigue and to anticipate when symptoms will worsen again.

To help people manage their fatigue, assessment and treatment approaches need to encompass the daily fluctuations and their interaction over time with activities of daily living.

Ecological momentary assessment (EMA) is a well-established method for capturing everyday experiences, including thoughts and behaviors, in their immediate context. As they go about their everyday lives, respondents are prompted multiple times a day, on a mobile device, to answer a brief set of questions about their momentary, "here and now", experience, e.g., "how happy are you right now?". On traditional self-report instruments, such as questionnaires, rating scales, and diaries, respondents are required to recall information or report on their beliefs and attitudes, which introduce risks of bias to the assessment attributable to memory limitations, personal beliefs, and self-perception. By sampling everyday experiences in real-time, EMA reduces these biases and errors.

The longitudinal nature of EMA even allows for assessment of dynamic processes and interactions that occur over short periods of time. Such fine-grained data are crucial for understanding how and why symptoms change during the day and to identify circumstances that may worsen or mitigate fatigue. This may lead to better treatment and symptom management.

A few studies in CP and ABI have demonstrated the feasibility and prospect of using EMA to capture the dynamics of fatigue. However, evidence is scarce regarding factors of everyday life that exacerbate or mitigate fatigue, although this information is essential for effective management strategies. Qualitative research indicates that several potential triggers of fatigue may be similar across CP and ABI.

Primary Objective:

1. To identify patterns of fatigue and antecedents of symptom exacerbation in daily life of adults with CP and ABI.

   Secondary Objectives:
2. To compare the dynamics of fatigue across CP, ABI, and neurotypical controls.
3. To identify factors in daily life that correlate with exacerbating fatigue symptoms.
4. To explore how physical activity, rest, and sleep influence fatigue patterns.

Design: We will use an intensive longitudinal observational study design. Participants will be asked to monitor in real-time for seven consecutive days. Notifications will pop up on their smartphone 10 times a day, and participants will be prompted to answer a brief survey about "how they are doing", "what they are doing", "where they are", and "who they are with", when they received the notification.

Participants will wear an accelerometer on their least affected thigh, and they will be asked to complete a sleep diary every morning in the seven-day period. The day prior to real-time monitoring, participants will meet with a research assistant to be instructed in the EMA protocol.

One week after real-time monitoring, participants will be invited to a feedback session, where the results of real-time monitoring of fatigue, activity, and sleep will be presented and discussed.

We will compare three groups of participants: Adults with CP, adults with ABI, and healthy volunteers without neurological conditions.

Participants with CP will be recruited via a public online announcement on the Elsass Foundation's website.

Participants with ABI will be recruited via two specialised brain injury rehabilitation centers (Vejlefjord Rehabilitering and Center for Rehabilitation of Brain Injury).

Healthy volunteers for the control group were initially planned to be recruited via the social network of the participants with CP or ABI. From August 2025, recruitment will be advertised publicly through social media platforms of the Neurorehabilitation Research and Knowledge Centre, Copenhagen University Hospital - Rigshospitalet (including newsletter, LinkedIn, and announcement on the webpage). The call for healthy volunteers will also be promoted through advocacy organizations for individuals with cerebral palsy or acquired brain injury, e.g., via social media platforms or their websites.

ELIGIBILITY:
Inclusion Criteria:

* Score of minimum 4 on the 7-item Fatigue Severity Scale (CP and ABI only)
* Speak, read, and write Danish
* Living in a private residence (i.e., not in institutional care or facilities providing 24-hour assistance)
* Able to walk independently or with assistive devices over short distances
* Able to operate a smartphone independently

Additional inclusion criteria for CP specifically:

* Self-reported diagnosis of CP
* Gross Motor Function Classification System (GMFCS) level ≤ II
* Communication Function Classification System level ≤ II

Additional inclusion criteria for ABI specifically:

* Self-reported diagnosis of ABI, including stroke, traumatic brain injury, brain infections, toxins, anoxia, or encephalopathy (transient ischemic attack, concussion or post-concussion syndrome, intracranial tumors, or progressive brain diseases are not included)
* Between three months and two years post-injury
* modified Rankin Scale (mRS) score ≤ 3

Exclusion Criteria:

* History of other neurological disorders or chronic fatigue syndrome requiring treatment
* Current substance or alcohol abuse
* Night shift work or travel across time zones (1 to 3 zones within the last week or 4 to 6 zones within the last two weeks or at least 7 zones within the last 4 weeks)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be residing in Denmark. Participants with CP will be recruited nationally via two sites located in the eastern and western part of Denmark, respectively: Glostrup and Kolding. They are not required to have any affiliation with clinical settings or organizations.
  Healthy volunteers will be recruited via a single site in the eastern part of Denmark (Glostrup).
  Participants with ABI will be recruited via two specialized rehabilitation centers in the eastern and western part of Denmark:
  1. Vejlefjord Rehabilitation, providing both inpatient and outpatient rehabilitation programs for children and adults with functional impairments following brain injury.
  2. Center for Rehabilitation of Brain Injury, providing outpatient rehabilitation services for individuals with acquired brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Ecological Momentary Assessment: "Fatigue item" | 10 times a day over 7 consecutive days
  A single item variable: "How tired do you feel right now?" Rated on an 11-point slider scale ranging from 0 (no fatigue) to 10 (severe fatigue).

SECONDARY OUTCOMES:
SENS motion® activity sensor | 7 consecutive days
  SENS motion® wearable activity sensor is an accelerometer that will be attached to the thigh using a patch. The accelerometer will be used to measure physical activity, sedentary behavior, and sleep. If the participants have any physical impairments, the patch will be worn on the least affected thigh.
Consensus Sleep Diary (CSD) | 1 time a day over 7 consecutive days
  The Consensus Sleep Diary (CSD) is a self-report 9-item instrument designed to track sleep patterns on a daily basis for typically 1-2 weeks. The questions ask about: (1) the time of getting into bed; (2) the time at which the individual attempted to fall asleep; (3) sleep onset latency; (4) number of awakenings; (5) duration of awakenings; (6) time of final awakening; (7) final rise time; (8) perceived sleep quality, rated on a 5-level scale from 1 (very poor) to 5 (very good); and (9) an additional space for open-ended comments from the respondent.
  We added two items from the expanded CSD for Morning about napping or dozing during the day: (10) number of naps/dozings; and (11) duration of naps/dozings.
  Participants are instructed to complete the CSD within one hour of getting out of bed in the morning.
Ecological Momentary Assessment "Energy item" | 10 times a day over 7 consecutive days
  A single item variable: "How much energy do you have right now?" Rated on an 11-point slider scale ranging from 0 (pictogram of an empty battery) to 10 (pictogram of a full battery).
Ecological Momentary Assessment: "Fatigue domain item" | 10 times a day over 7 consecutive days
  A single item variable: "How does your fatigue feel right now?" Response categories are: "Primarily physical", "Primarily mental", "Both", "Neither", and "Not relevant"
Ecological Monetary Assessment: "Alert item" | 10 times a day over 7 consecutive days
  A single item variable: "How alert do you feel right now?". Rated on an 11-point slider scale ranging from 0 (not at all) to 10 (very much).
Ecological Momentary Assessment "Exhaustion item" | 10 times a day over 7 consecutive days
  A single item variable: "How exhausted do you feel right now?" Rated on an 11-point slider scale ranging from 0 (not at all) to 10 (very much).
Ecological Momentary Assessment "Pain item" | 10 times a day over 7 consecutive days
  A single item variable: "How much pain do you have right now?" Rated on an 11-point slider scale ranging from 0 (no pain) to 10 (worst pain imaginable).
Ecological Momentary Assessment "Sleepy item" | 10 times a day over 7 consecutive days
  A single item variable: "How sleepy do you feel right now?" Rated on an 11-point slider scale ranging from 0 (not at all) to 10 (very much)
Ecological Momentary Assessment: "Concentration item" | 10 times a day over 7 consecutive days
  A single item variable: "How well are you able to concentrate right now?" Rated on an 11-point slider scale ranging from 0 (not at all) to 10 (very much).
Ecological Momentary Assessment: "Effort item" | 10 times a day over 7 consecutive days
  A single item variable: "How much of an effort is it to do anything right now?" Rated on an 11-point slider scale ranging from 0 (none at all) to 10 (very much).
Ecological Momentary Assessment: "Happiness item" | 10 times a day over 7 consecutive days
  A single item variable: "How happy do you feel right now?" Rated on an 11-point slider scale ranging from 0 (not at all) to 10 (very much).
Ecological Momentary Assessment: "Sadness item" | 10 times a day over 7 consecutive days
  A single item variable: "How sad do you feel right now?" Rated on an 11-point slider scale ranging from 0 (not at all) to 10 (very much).
Ecological Momentary Assessment: "Anxious item" | 10 times a day over 7 consecutive days
  A single item variable: "How anxious do you feel right now?" Rated on an 11-point slider scale ranging from 0 (not at all) to 10 (very much).
Ecological Momentary Assessment: "Irritability item" | 10 times a day over 7 consecutive days
  A single item variable: "How irritable do you feel right now?" Rated on an 11-point slider scale ranging from 0 (not at all) to 10 (very much).
Ecological Momentary Assessment: "Activity item" | 10 times a day over 7 consecutive days
  A single item variable: "What were you doing when you received the notification?" Multiple choice response.
Ecological Momentary Assessment: "Physical demand item" | 10 times a day over 7 consecutive days
  A single item variable: "How physically demanding is the task you were doing?" Rated on an 11-point slider scale ranging from 0 (not at all) to 10 (very much).
Ecological Momentary Assessment: "Mental demand item" | 10 times a day over 7 consecutive days
  A single item variable: "How mentally demanding is the task you were doing?" Rated on an 11-point slider scale ranging from 0 (not at all) to 10 (very much).
Ecological Momentary Assessment: "Motivation item" | 10 times a day over 7 consecutive days
  A single item variable: "How motivated were you for the task you were doing?" Rated on an 11-point slider scale ranging from 0 (not at all) to 10 (very much).
Ecological Momentary Assessment: "Location item" | 10 times a day over 7 consecutive days
  A single item variable: "Where were you when you received the notification?" Multiple choice response.
Ecological Momentary Assessment: "Sensory load item" | 10 times a day over 7 consecutive days
  A single item variable: "How many sensory impressions were present around you when you received the notification?" Rated on a 5-point Likert-type scale: 0 (Very low degree), 1 (Low degree), 2 (Some degree), 3 (High degree), and 4 (Very high degree).
Ecological Momentary Assessment: "Company item" | 10 times a day over 7 consecutive days
  A single item variable: "Who were with you when you received the notification?" Multiple choice response.

OTHER OUTCOMES:
Fatigue Severity Scale (FSS) | Baseline
  A self-report 9-item questionnaire measuring the impact of fatigue in daily life. The scale provides a total average score of the nine items, ranging from 1 to 7, with 1 indicating no or little experience with functional limitations due to fatigue and 7 indicating severe functional limitations due to fatigue.
The Fatigue Impact and Severity Self-Asssessment (FISSA) | Baseline
  A self-administered 37-item questionnaire. It includes a total fatigue score (the sum of items 1-31), ranging from 31 (low fatigue) to 157 (high fatigue), and two subscales: The Impact Subscale (items 1-17, score range from 17 to 87) and the Management and Activity Modification Subscale (items 18-31, score range from 14 to 70). Higher scores indicate more fatigue. The last 6 items (items 32-37) are a mix of multiple choice and open-ended questions investigating daily fatigue and management that are not included in any scores.
  The complete FISSA will be administered to participants with cerebral palsy only. The last 6 items will also be administered to participants with acquired brain injury.
Dutch Multifactor Fatigue Scale (DMFS) | Baseline
  The Dutch Multifactor Fatigue Scale (DMFS) is a self-administered questionnaire designed to assess the multidimensional nature of fatigue and coping strategies in individuals with acquired brain injury.
  DMFS has 38 items scored on a 5-point Likert-type scale ranging from 1 (No, I strongly disagree) to 5 (Yes, I strongly agree). DMFS includes 5 subscales: Impact of Fatigue (score range from 11 to 55), Signs and Direct Consequences of Fatigue (score range from 9 to 45), Mental Fatigue (score range from 7 to 35), Physical Fatigue (score range from 6 to 30), and Coping with Fatigue (score range from 5 to 25). Higher scores indicate more fatigue or worse coping with fatigue.
  DMFS will be administered to participants with acquired brain injury only.
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  A self-report questionnaire assessing sleep quality over a one-month period. The questionnaire includes 19 self-rated questions and 5 questions rated by the bed partner or roommate, covering different sleep-related factors such as bedtime habits, sleep disturbances, sleep duration, and daytime impairments. The 19 self-rated items are scored from 0 to 3 to create seven component scores, which are added to produce a global PSQI score, ranging from 0 (no difficulty) to 21 (severe difficulty).
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  A 9-item self-report questionnaire to screen for depression. Each question is scored on a scale from 0 to 3 with higher scores indicating more severe symptoms.
Perceived Stress Scale (PSS) | Baseline
  A self-report 10-item questionnaire designed to measure psychological stress. Items are scored on a scale from 0 to 4. Higher scores indicate more perceived stress.
EuroQol 5-Dimension Health Questionnaire 5 Level (EQ-5D-5L) | Baseline
  The EQ-5D-5L is a standardized instrument for measuring health-related quality of life. It contains the EQ-5D-5L Descriptive System and the EQ Visual Analog Scale (EQ VAS). The descriptive system comprises 5 dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, and Anxiety/depression. Each dimension is rated on five levels: 1 (No problems), 2 (Slight problems), 3 (Moderate problems), 4 (Severe problems), and 5 (Extreme problems). The ratings on the five dimensions define a health profile. Health profiles will be converted to health state index scores using the Danish EQ-5D-5L value set, which ranges from -0.757 (worst health) to 1 (perfect health).
  The EQ VAS records the respondent's self-rated health on a vertical, visual analog scale, ranging from 0-100, where the endpoints are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0).
WHODAS-12 | Baseline
  A short, self-administered questionnaire developed by the World Health Organisation to measure disability and functioning covering mobility, cognition, activities of daily living, participation in society and getting along with others. Items are scored on a 5-point Likert scale from 0 to 4 with higher scores indicating higher disability.
Physical Activity Scale 2 (PAS2) | Baseline
  The Physical Activity Scale (PAS2) is a self-administered 9-item questionnaire that assesses physical activity. Respondents estimate daily hours and minutes spent on (1) sleeping, (2) sedentary work, (3) standing or walking work, (4) heavy physical work, (5) riding a bicycle or walking for transportation to and from work, and (6) sedentary activities during leisure time. In addition, respondents estimate weekly hours and minutes of (7) light, (8) moderate, and (9) vigorous physical activity during leisure time. The item responses are summarised as average time spent per day on sedentary behavior, light physical activity, moderate physical activity, and vigorous physical activity.
Montreal Cognitive Asessment (MoCA) | Baseline
  A brief screening tool to detect mild cognitive impairment. The Montreal Cognitive Assessment is scored out of a total of 30 points. A score of 26 or above is considered normal, while scores below 26 may indicate mild cognitive impairment. Scores can be used to indicate severity: 18-25 indicates mild impairment, 10-17 indicates moderate impairment, and below 10 indicates severe impairment.
The Hearts Test, subtest from Oxford Cognitive Screen | Baseline
  Assessment of visual attention and spatial processing. The total time taken for the task is recorded and 1 point is given for every correctly cancelled heart shape. The overall accuracy is recorded as "Total Correct" (maximum score = 50). This score contributes to the overall assessment of attention, and reflects performance of sustained and selected attention. A space asymmetry score is calculated, and a positive score indicates left-sided egocentric neglect, and a negative score indicates right-sided egocentric neglect. An object asymmetry score is calculated, and a positive value indicates left allocentric neglect. A negative asymmetry score indicates right allocentric neglect.
6 minute walk test | Baseline
  A standardised assessment of functional exercise capacity.
Background information: Gender | Baseline
  Self-reported. Single choice from 4 response options.
Background information: Ethnicity | Baseline
  Self-reported. 3 response options.
Background information: Current Employment | Baseline
  Employment status is self-reported using 11 predefined response options. If currently employed, respondents indicate the average number of working hours per week. If on sick leave, respondents report their employment status prior to taking leave. If currently studying, respondents specify the type of education they are enrolled in.
Background information: Educational level | Baseline
  The highest completed level of eduction is self-reported using 11 response options.
Background information: Marital status | Baseline
  Self-reported. 4 response options
Background information: Housing situation | Baseline
  Respondents report their current living arrangement using six predefined reponse options. These options capture whether they live alone or with others, and whether they reside in their own home or in a shared living arrangement, with either a private or shared room.
Background information: Household composition | Baseline
  Respondents report the number of people they currently live with and identify their relationship to these individuals by selecting from seven predefined categories: Partner, children under 25 years old, children above 25 years old, parents, other family members, friends or other types of relationships, and other.
Background information: Body Mass Index (BMI) | Baseline
  BMI is calculated based on self-reported weight in kilograms and height in meters and centimeters.
Background information: Tobacco and nicotine use | Baseline
  Respondents indicate whether and how frequently they use tobacco or nicotine products using a five-point scale. If any use is reported, respondents select the type(s) of product used from five predefined categories. If cigarette use is indicated, the average number of cigarettes smoked per day is reported.
Background information: Alcohol consumption | Baseline
  The average number of standard drinks consumed per week is self-reported.
Background information: Use of other substances | Baseline
  Respondents indicate their use of substances other than alcohol or nicotine using four predefined response categories. If any use is reported, respondents may specify the type of substances used in an open-text field.
Background information: Physical or mental diseases | Baseline
  Respondents specify any illness, diagnosis, handicap, or symptoms using an open-text field.
Background information: Medicine use | Baseline
  Respondents indicate their current use of medication by selecting one of four predefined response options: "No", "As needed", "Regularly", or "Prefer not to answer". If any use is reported, respondents specify the type(s) of medication used by selecting from 14 predefined categories. For each category selected, they are asked to name the specific medication(s) taken, and report the frequency and duration of use. Respondents are also asked to indicate any adverse effects.
Background Information: Smartphone use | Baseline
  An 8-item self-report questionnaire covering smartphone usage and habits. Respondents indicate whether they own a smartphone, how frequently they use it, and for what purposes. They also report where their smartphone is typically located when at home, at work or during study, and while in transit. Additionally, respondents indicate whether they use their smartphone to monitor their health and, if so, which health-related apps they have used.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Norup, Ph.D., Study Director — Neurorehabilitation Research and Knowledge Centre, Rigshospitalet
Locations (1):
- Neurorehabilitation Research and Knowledge Centre, Rigshospitalet, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided